CLINICAL TRIAL: NCT00218075
Title: Behavioral Strategies to Maximize the Efficacy of Pharmacotherapy for Cocaine Dependence: Relapse Prevention With Contingency Management Procedures
Brief Title: Behavioral Therapy Combined With Carbidopa/Levodopa for the Treatment of Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Texas (Other)
Responsible Party: Principal Investigator, Joy Schmitz, Professor - Psy, Behavioral Science, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09262-9; P50DA009262 (NIH); P50-09262-9; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Cocaine Abuse; Cocaine-Related Disorders
Keywords: Cocaine addiction; cocaine treatment
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Levodopa; Carbidopa; Secondary Prevention

INTERVENTIONS:
Drug: Levodopa
Drug: Carbidopa
Behavioral: Clinical Management
Behavioral: Relapse Prevention Therapy
Behavioral: Contingency Management

SUMMARY:
Cocaine dependence is a major public health problem; an effective primary treatment for cocaine dependent individuals has yet to be found. The purpose of this study is to examine the effectiveness of levodopa and carbidopa in treating cocaine dependent individuals. In addition, this study will examine the effects of incentive rewards for treatment compliance.

DETAILED DESCRIPTION:
Cocaine is a strong central nervous system stimulant that is widely abused throughout the United States. Due to its widespread use, it is important to develop an effective treatment for cocaine dependence. Levodopa is a medication that is used alone or in combination with carbidopa to treat Parkinson's disease. The purpose of this study is to determine the possible interactions between behavioral interventions and carbidopa/levodopa in order to treat cocaine dependent individuals.

This study will last 12 weeks and will involve two phases. The first phase will include three therapy conditions: 1) clinical management only, 2) clinical management and relapse prevention therapy, and 3) clinical management, relapse prevention therapy, and contingency management. All of the conditions in the first phase will be evaluated incrementally under active and placebo conditions while participants receive carbidopa/levodopa.

The second phase of the study will examine the contingency management procedure applications. Each of the three contingency management procedure applications targets specific behaviors that, when reinforced, may interact with carbidopa/levodopa to produce clinical benefits. Participants will receive relapse prevention therapy combined with a contingency management procedure that targets clinic attendance, medication compliance, and cocaine abstinence. Study visits will occur weekly throughout the study. In addition, participants will complete a one-year follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current cocaine dependence
* Provides at least one positive urine test for cocaine during study screening
* Good general health, based on a physical exam, lab tests, and an electrocardiogram
* Reads and writes English at a sixth grade level

Exclusion Criteria:

* Current Axis I depressive, psychotic, or anxiety disorder
* Currently in jail
* Pregnant or breastfeeding
* Requires certain medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 2000-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Cocaine use

SECONDARY OUTCOMES:
Medication compliance
treatment retention
severity of addiction-related problems

CONTACTS AND LOCATIONS:
Overall Officials: John Grabowski, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States